CLINICAL TRIAL: NCT04608916
Title: Efficacy of Surgical Diathermy in Eradicating Cutibacterium Acnes From Surgical Skin Incision During Shoulder Arthroplasty
Acronym: Electrocautery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, H. Mike Kim, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MU IRB 2020
Record Dates: First submitted 2020-10-25; First posted 2020-10-29 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Infection, Bacterial
Keywords: Shoulder arthroplasty; Infection; Periprosthetic joint infection; Cutibaterium acnes; Diathermy; Electrocautery
MeSH Terms: conditions — Bacterial Infections; Infections; Fever

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scalpel incision group (Active Comparator): This group of patients will receive skin incision made with use of a scalpel blade.
  Interventions: Procedure: Using scalpel blade to make skin incision
- Electrocautery incision group (Experimental): This group of patients will receive skin incision made with use of electrocautery.
  Interventions: Procedure: Using surgical diathermy to make skin incision

INTERVENTIONS:
Procedure: Using surgical diathermy to make skin incision — Using surgical diathermy to make skin incision during shoulder arthroplasty
  Arms: Electrocautery incision group
Procedure: Using scalpel blade to make skin incision — Using scaple blade to make skin incision during shoulder arthroplasty
  Arms: Scalpel incision group

SUMMARY:
Periprosthetic infection following shoulder arthroplasty is a devastating complication. Diagnosing and treating periprosthetic shoulder infection poses a significant challenge. At the forefront of this issue is Cutibacterium acnes because the current prophylactic regimens are insufficient to eradicate C acnes from the surgical field. It is believed that C acnes infections occur during surgery when the sebaceous glands in the skin are cut and exposed, leading to C acnes contaminating the surgeon's instruments and gloves and, thus, the surgical wound. The purpose of this study is to examine if making skin incisions using electrocautery will result in decreased C acnes contamination during shoulder arthroplasty. To this end, we propose a randomized clinical trial where patients undergoing shoulder arthroplasty are randomized into two groups - Electrocautery incision group (Electro) vs. Scalpel incision group (Scalpel) - and swab cultures are obtained from the skin incision and operating surgeon's gloves and forceps

DETAILED DESCRIPTION:
Periprosthetic infection following shoulder arthroplasty is a devastating complication. Infected shoulder arthroplasty not only causes an unexpected health hazard to patients but also imposes a heavy financial burden at both individual and societal levels. The rates of periprosthetic shoulder infection (PSI) have been reported to be 0.80% to 1.46%, but the number of infections is likely to increase as shoulder arthroplasty becomes more commonplace in an aging active population. Diagnosing and treating PSI poses a significant challenge. Unlike periprosthetic infection in other joints, PSI lacks the typical clinical signs and laboratory findings of infection due to the indolent nature of the offending pathogens. At the forefront of this issue is Cutibacterium acnes. Although the typical Staphylococcus, Streptococcus, and Corynebacterium species that reside on the skin surface are the primary targets of most surgical infection prophylaxis regimens, C acnes has emerged as a problematic bacterium because the current prophylactic regimens are insufficient to eradicate C acnes from the surgical field.

C acnes is one of the most common pathogens of infections after shoulder surgery. It is a commensal, gram-positive anaerobic bacillus that resides in the sebaceous glands associated with hair follicles. The colonization with C acnes of the front and back side of the shoulder epidermis is greater than that of other regions of the body because of the high density of the sebaceous glands in that area. C acnes can cause low-grade infections after shoulder surgery, and it has been shown that it is the most commonly detected bacterium after revision shoulder arthroplasty surgery. During revision shoulder arthroscopy cases performed for pain, stiffness, or weakness, 30% of patients had positive culture findings, and 80% of those findings were positive for C acnes. It is believed that C acnes infections occur during surgery when the sebaceous glands in the skin are cut and exposed, leading to C acnes contaminating the surgeon's instruments and gloves and, thus, the surgical wound. Recent studies showed that hydrogen peroxide and benzoyl peroxide were more effective than the conventional skin preparation methods in decreasing the C acnes load in the skin, but as high as 17% of the cultures were still positive for C acnes even with these new measures. Thus, despite all the efforts to eradicate C acnes from the shoulder, C acnes remain an elusive pathogen that is potentially contaminating tens of thousands of shoulder arthroplasties each year.

Surgical diathermy (or electrocautery) has been used routinely for tissue dissection and hemostasis during surgical procedures. In the cutting mode, the use of an electrode delivering a pure continuous sinusoidal wave of low voltage produces as high temperatures as 1000℃, which heats cells within the tissue so rapidly that they vaporize, leaving a cavity within the cell matrix. The heat created dissipates as a stream rather than being transmitted into adjacent tissues. This allows tissue cleavage without damage to surrounding areas. The electrode does not need to be in contact with tissue as an arc is formed producing a clean cut. With the coagulation mode on high power, cutting also occurs, but this produces a larger zone of greater thermal damage. Electrocautery can be used for dissecting fascia and muscle layers, as well as achieving hemostasis, and it has become an integral part of modern surgical practice. A number of clinical studies evaluated the safety and efficacy of cutting electrocautery for surgical incisions in general, plastic, otorhinolaryngological, orthopedic, neurosurgical, and gynecologic procedures. Additionally, systematic reviews and meta-analyses were conducted for the same purposes. The majority of these studies showed that using electrocautery to cut the skin provided the benefits of reduced bleeding, a quicker incision, and decreased postoperative pain with no increase of wound complications when compared to scalpel incisions. Given the high temperatures generated at the tip of an electrode of electrocautery, it is reasonable to assume that making a skin incision with electrocautery could potentially destroy exposed colonies of C acnes in hair follicles and sebaceous glands open on the incisional surface of the skin. The purpose of this study is to examine if making skin incisions using electrocautery will result in decreased C acnes contamination during shoulder arthroplasty. To this end, we propose a randomized clinical trial where patients undergoing shoulder arthroplasty are randomized into two groups - Electrocautery incision group (Electro) vs. Scalpel incision group (Scalpel) - and swab cultures are obtained from the skin incision and operating surgeon's gloves and forceps.

ELIGIBILITY:
Inclusion Criteria:

* Adult male patients (>18 years old) who undergo primary shoulder arthroplasty (either anatomic or reverse shoulder arthroplasty)

Exclusion Criteria:

* History of ipsilateral shoulder postoperative infection
* Administration of any antibiotics within a month prior to the index procedure
* Active acne at the surgical site
* History of psoriatic or eczematous lesions about the shoulder area
* Revision arthroplasty cases
* Minors (< 18 years old)
* Female patients
* Prisoners
* Patients who cannot understand English enough to give an informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Proportions of positive C acnes cultures | 2 weeks following surgery
  Proportions of positive C acnes cultures

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD with other researchers

REFERENCES:
- [Background] Padegimas EM, Maltenfort M, Ramsey ML, Williams GR, Parvizi J, Namdari S. Periprosthetic shoulder infection in the United States: incidence and economic burden. J Shoulder Elbow Surg. 2015 May;24(5):741-6. doi: 10.1016/j.jse.2014.11.044. Epub 2015 Jan 13. PMID 25595360
- [Background] van Diek FM, Pruijn N, Spijkers KM, Mulder B, Kosse NM, Dorrestijn O. The presence of Cutibacterium acnes on the skin of the shoulder after the use of benzoyl peroxide: a placebo-controlled, double-blinded, randomized trial. J Shoulder Elbow Surg. 2020 Apr;29(4):768-774. doi: 10.1016/j.jse.2019.11.027. PMID 32197765
- [Background] Foruria AM, Fox TJ, Sperling JW, Cofield RH. Clinical meaning of unexpected positive cultures (UPC) in revision shoulder arthroplasty. J Shoulder Elbow Surg. 2013 May;22(5):620-7. doi: 10.1016/j.jse.2012.07.017. Epub 2012 Sep 13. PMID 22981448
- [Background] Achermann Y, Sahin F, Schwyzer HK, Kolling C, Wust J, Vogt M. Characteristics and outcome of 16 periprosthetic shoulder joint infections. Infection. 2013 Jun;41(3):613-20. doi: 10.1007/s15010-012-0360-4. Epub 2012 Nov 3. PMID 23124880
- [Background] Horneff JG 3rd, Hsu JE, Voleti PB, O'Donnell J, Huffman GR. Propionibacterium acnes infection in shoulder arthroscopy patients with postoperative pain. J Shoulder Elbow Surg. 2015 Jun;24(6):838-43. doi: 10.1016/j.jse.2015.03.008. PMID 25979553
- [Background] Falconer TM, Baba M, Kruse LM, Dorrestijn O, Donaldson MJ, Smith MM, Figtree MC, Hudson BJ, Cass B, Young AA. Contamination of the Surgical Field with Propionibacterium acnes in Primary Shoulder Arthroplasty. J Bone Joint Surg Am. 2016 Oct 19;98(20):1722-1728. doi: 10.2106/JBJS.15.01133. PMID 27869623
- [Background] Ly J, Mittal A, Windsor J. Systematic review and meta-analysis of cutting diathermy versus scalpel for skin incision. Br J Surg. 2012 May;99(5):613-20. doi: 10.1002/bjs.8708. Epub 2012 Feb 24. PMID 22367850
- [Background] Ismail A, Abushouk AI, Elmaraezy A, Menshawy A, Menshawy E, Ismail M, Samir E, Khaled A, Zakarya H, El-Tonoby A, Ghanem E. Cutting electrocautery versus scalpel for surgical incisions: a systematic review and meta-analysis. J Surg Res. 2017 Dec;220:147-163. doi: 10.1016/j.jss.2017.06.093. Epub 2017 Jul 26. PMID 29180177
- [Background] Kearns SR, Connolly EM, McNally S, McNamara DA, Deasy J. Randomized clinical trial of diathermy versus scalpel incision in elective midline laparotomy. Br J Surg. 2001 Jan;88(1):41-4. doi: 10.1046/j.1365-2168.2001.01625.x. PMID 11136307
- [Background] Hemsell DL, Hemsell PG, Nobles B, Johnson ER, Little BB, Heard M. Abdominal wound problems after hysterectomy with electrocautery vs. scalpel subcutaneous incision. Infect Dis Obstet Gynecol. 1993;1(1):27-31. doi: 10.1155/S1064744993000079. PMID 18476202